CLINICAL TRIAL: NCT01538043
Title: Spa Therapy in Knee Osteoarthritis: Study on Cost/Effectiveness - Cost/Utility and Possible Mechanisms of Action
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, fioravanti antonella, medical doctor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAC2010
Record Dates: First submitted 2012-02-13; First posted 2012-02-23 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Cost-effectiveness analysis; Cost-utility analysis; Osteoarthritis; Spa therapy; Randomized clinical trial; Mechanisms of action
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Balneology; Mud Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- local mud packs and thermal-mineral bath (Active Comparator): 50 patients with primary knee OA will be treated with daily local mud packs and thermal-mineral bath at Chianciano Terme Spa Center (Siena, Italy) for a total of 12 applications carried out over a period of two weeks
  Interventions: Other: local mud-pack therapy and balneotherapy
- regular routine ambulatory care (No Intervention): 50 patients, the control group, will continue regular routine ambulatory care

INTERVENTIONS:
Other: local mud-pack therapy and balneotherapy — local mud-pack therapy and thermal-mineral bath at Chianciano Terme Spa Center (Siena, Italy) for a total of 12 applications carried out over a period of two weeks
  Other Names: mud pack therapy
  Arms: local mud packs and thermal-mineral bath

SUMMARY:
The aim of this study is to evaluate both cost/effectiveness- cost/utility and the possible mechanisms of action of spa therapy in patients with primary knee osteoarthritis (OA).

DETAILED DESCRIPTION:
OA is the most common rheumatic disease and the most important from the social-economic point of view because of its frequency, causing functional impairment and disability in older people, important health resource utilization and costs (drugs, physical therapies, spa therapy, surgical prothesis, early retirement).

Thermal therapy is one of the most commonly used non-pharmacological approaches for OA, but it is still being discussed and its role in modern medicine is still not clear. The action mechanisms of mud packs and thermal baths are not completely known, and it is difficult to distinguish the effects of thermal applications from the benefits that could be derived from a stay in a spa environment. Furthermore, there are no data about cost analysis of spa therapy in OA.

The aim of this study is to analyze for the first time the cost/effectiveness- cost/utility for spa therapy in comparison to conventional treatments in knee OA (one-year-follow-up)and to assess changes of some biomarkers or mediators of cartilage damage in order to identify new possible mechanisms of action of spa therapy in rheumatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from OA of the knee according to American College of Rheumatology (ACR) criteria and to standard radiography of the knee

Exclusion Criteria:

* patients enrolled in other research protocols
* patients that have been treated with mud-pack therapy and balneotherapy in the last 9 months
* patients affected by neoplastic diseases or in the last five years, with cardiovascular disease of recent onset, suffering from inflammatory diseases in the acute phase, serious impairment of hematopoietic, renal and hepatic systems, other inflammatory rheumatic or autoimmune disorders, or unable to complete the questionnaires and the daily diary for the collection of socio-economic data

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
cost/effectiveness- cost/utility for spa therapy compared to conventional treatments in knee osteoarthritis | baseline and twelve months
  to evaluate for the first time cost/effectiveness- cost/utility for spa therapy compared to conventional treatments by a randomized single blind controlled trial in knee osteoarthritis

SECONDARY OUTCOMES:
changes of certain markers or mediators of cartilage damage | baseline and two weeks
  to assess changes of certain markers or mediators of cartilage damage in order to identify new possible mechanisms of action of spa therapy in rheumatic diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Fioravanti, MD, Principal Investigator — Rheumatology Unit- Azienda Ospedaliera Universitaria Senese- Siena- Italy
Locations (1):
- Rheumatology Unit Azienda Ospedaliera Universitaria Senese, Siena, Italy

REFERENCES:
- [Background] Fioravanti A, Valenti M, Altobelli E, Di Orio F, Nappi G, Crisanti A, Cantarini L, Marcolongo R. Clinical efficacy and cost-effectiveness evidence of spa therapy in osteoarthritis. The results of "Naiade" Italian Project. Panminerva Med. 2003 Sep;45(3):211-7. PMID 14618120
- [Background] Cantarini L, Leo G, Giannitti C, Cevenini G, Barberini P, Fioravanti A. Therapeutic effect of spa therapy and short wave therapy in knee osteoarthritis: a randomized, single blind, controlled trial. Rheumatol Int. 2007 Apr;27(6):523-9. doi: 10.1007/s00296-006-0266-5. Epub 2006 Nov 15. PMID 17106661
- [Background] Fioravanti A, Iacoponi F, Bellisai B, Cantarini L, Galeazzi M. Short- and long-term effects of spa therapy in knee osteoarthritis. Am J Phys Med Rehabil. 2010 Feb;89(2):125-32. doi: 10.1097/PHM.0b013e3181c1eb81. PMID 19884812
- [Background] Fioravanti A, Cantarini L, Bacarelli MR, de Lalla A, Ceccatelli L, Blardi P. Effects of spa therapy on serum leptin and adiponectin levels in patients with knee osteoarthritis. Rheumatol Int. 2011 Jul;31(7):879-82. doi: 10.1007/s00296-010-1401-x. Epub 2010 Mar 18. PMID 20237929
- [Background] Fioravanti A, Cantarini L, Guidelli GM, Galeazzi M. Mechanisms of action of spa therapies in rheumatic diseases: what scientific evidence is there? Rheumatol Int. 2011 Jan;31(1):1-8. doi: 10.1007/s00296-010-1628-6. Epub 2010 Dec 1. PMID 21120502
- [Background] Fioravanti A, Giannitti C, Bellisai B, Iacoponi F, Galeazzi M. Efficacy of balneotherapy on pain, function and quality of life in patients with osteoarthritis of the knee. Int J Biometeorol. 2012 Jul;56(4):583-90. doi: 10.1007/s00484-011-0447-0. Epub 2011 May 15. PMID 21573819
- [Background] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131
- [Derived] Ciani O, Pascarelli NA, Giannitti C, Galeazzi M, Meregaglia M, Fattore G, Fioravanti A. Mud-Bath Therapy in Addition to Usual Care in Bilateral Knee Osteoarthritis: An Economic Evaluation Alongside a Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2017 Jul;69(7):966-972. doi: 10.1002/acr.23116. Epub 2017 Jun 7. PMID 27723261
- [Derived] Chung KC, Kotsis SV, Burns PB, Burke FD, Wilgis EFS, Fox DA, Kim HM. Seven-Year Outcomes of the Silicone Arthroplasty in Rheumatoid Arthritis Prospective Cohort Study. Arthritis Care Res (Hoboken). 2017 Jul;69(7):973-981. doi: 10.1002/acr.23105. Epub 2017 Jun 9. PMID 27696739
- [Derived] Fioravanti A, Giannitti C, Cheleschi S, Simpatico A, Pascarelli NA, Galeazzi M. Circulating levels of adiponectin, resistin, and visfatin after mud-bath therapy in patients with bilateral knee osteoarthritis. Int J Biometeorol. 2015 Nov;59(11):1691-700. doi: 10.1007/s00484-015-0977-y. Epub 2015 Mar 7. PMID 25750093